CLINICAL TRIAL: NCT01464931
Title: An Open-label Study to Evaluate the Safety of Multiple Doses of Denosumab 120 mg Administered Subcutaneously in Subjects With Severe Chronic Kidney Disease (CKD) and CKD on Dialysis
Brief Title: Multiple Dose Study to Evaluate the Safety of Multiple Doses of Denosumab 120 mg in Adults With Severe Chronic Kidney Disease (CKD) and CKD on Dialysis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20101361
Record Dates: First submitted 2011-10-17; First posted 2011-11-04 (Estimated); Results first posted 2016-02-19 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-01

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Denosumab (Experimental): Participants received two 120 mg doses of denosumab administered subcutaneously on Day 1 and Day 29.
  Interventions: Drug: Denosumab

INTERVENTIONS:
Drug: Denosumab — Adminstered by subcutaneous injection
  Other Names: XGEVA; AMG 162

SUMMARY:
The primary objective was to evaluate the incidence of clinically significant hypocalcemia following multiple 120 mg subcutaneous doses of denosumab in patients with severe chronic kidney disease (CKD) and CKD on dialysis

ELIGIBILITY:
Inclusion Criteria:

* Subjects at least 18 years old with severe CKD (defined as creatinine clearance < 30 mL/min at both screening assessments) and CKD requiring hemodialysis
* Additional inclusion criteria apply

Exclusion Criteria:

* Subjects must have calcium, phosphate, and magnesium levels appropriate for their condition and must not have other uncontrolled co-morbidities.
* Additional exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-11; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (7):
- United States (7):
  - Research Site, Tempe, Arizona
  - Research Site, Denver, Colorado
  - Research Site, Pembroke Pines, Florida
  - Research Site, Meridian, Idaho
  - Research Site, Detroit, Michigan
  - Research Site, Orangeburg, South Carolina
  - Research Site, San Antonio, Texas

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Severe CKD: Participants with severe chronic kidney disease (CKD; defined as creatinine clearance < 30 mL/min) received two 120 mg doses of denosumab administered subcutaneously on Day 1 and Day 29.
- ESRD: Participants with end-stage renal disease (ESRD) requiring dialysis received two 120 mg doses of denosumab administered subcutaneously on Day 1 and Day 29.
Period: Overall Study
Arm/Group | Severe CKD | ESRD
Started | 16 | 16
Completed | 15 | 16
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Severe CKD | ESRD | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.2 (9.5) | 65.9 (12.4) | 72.5 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Significant Hypocalcemia
Description: Clinically significant hypocalcemia is defined as albumin-adjusted calcium < 7.0 mg/dL or symptomatic hypocalcemia. Symptomatic hypocalcemiais is defined as both a clinical adverse event of hypocalcemia and a concomitant symptom of hypocalcemia (e.g., hypoesthesia, paresthesia, muscle cramps, seizure, prolonged QT interval) that occurred along with the hypocalcemia event or decreased serum calcium levels.
Time Frame: 113 days
Population: Safety Analysis Set (all participants who received at least 1 dose of denosumab)
Measure: Number; unit: participants
Arm/Group | Severe CKD | ESRD
Number analyzed (Participants) | 16 | 16
participants | 1 | 2

2. Secondary Outcome: Number of Participants With Hypocalcemia Determined by CTCAE v.4.0 Criteria
Description: The severity of hypocalcemia (a low concentration of calcium, corrected for albumin, in the blood) was graded according to the common terminology criteria for adverse events (CTCAE) v.4.0 criteria: Grade 1: albumin-adjusted serum calcium < lower limit of normal (LLN; 9.2 mg/dL) to 8.0 mg/dL; Grade 2: albumin-adjusted serum calcium < 8.0 to 7.0 mg/dL; Grade 3: albumin-adjusted serum calcium < 7.0 to 6.0 mg/dL; Grade 4: albumin-adjusted serum calcium < 6.0 mg/dL.
Time Frame: 113 days
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | Severe CKD | ESRD
Number analyzed (Participants) | 16 | 16
participants
  Grade 1 | 12 | 6
  Grade 2 | 3 | 9
  Grade 3 | 0 | 1
  Grade 4 | 0 | 0

3. Secondary Outcome: Number of Participants With Hypophosphatemia Determined by CTCAE v.4.0 Criteria
Description: The severity of hypophosphatemia (a low concentration of phosphates in the blood) was graded according to the common terminology criteria for adverse events (CTCAE) v.4.0 criteria: Grade 1: < LLN (3 mg/dL) - 2.5 mg/dL; Grade 2: < 2.5 - 2.0 mg/dL; Grade 3: < 2.0 - 1.0 mg/dL; Grade 4: < 1.0 mg/dL.
Time Frame: 113 days
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | Severe CKD | ESRD
Number analyzed (Participants) | 16 | 16
participants
  Grade 1 | 0 | 0
  Grade 2 | 2 | 1
  Grade 3 | 0 | 5
  Grade 4 | 0 | 0

4. Secondary Outcome: Number of Participants With Hypomagnesemia Determined by CTCAE v.4.0 Criteria
Description: The severity of hypomagnesemia (a low concentration of magnesium in the blood) was graded according to the common terminology criteria for adverse events (CTCAE) v.4.0 criteria: Grade 1: < LLN (1.5 mg/dL) - 1.2 mg/dL; Grade 2: < 1.2 - 0.9 mg/dL; Grade 3: < 0.9 - 0.7 mg/dL; Grade 4: < 0.7 mg/dL.
Time Frame: 113 days
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | Severe CKD | ESRD
Number analyzed (Participants) | 16 | 16
participants
  Grade 1 | 2 | 0
  Grade 2 | 0 | 0
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0

5. Secondary Outcome: Percent Change From Baseline in Albumin-adjusted Serum Calcium Over Time
Time Frame: Baseline and Days 2, 3, 6, 8, 11, 15, 22, 29, 30, 31, 34, 36, 39, 43, 57, 71, 85, and 113
Population: Safety analysis set with available data at each time point
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Severe CKD | ESRD
Number analyzed (Participants) | 16 | 16
percent change
  Day 2 (N=16, 16) | -0.55 (3.56) [-1.28 to 0.51] | 1.21 (4.66) [-054 to 4.52]
  Day 3 (N=16, 16) | -3.20 (5.99) [-6.88 to 0.19] | -1.86 (5.82) [-7.11 to 2.38]
  Day 6 (N=16, 16) | -4.27 (7.42) [-7.77 to -0.90] | -7.34 (8.75) [-13.62 to 4.15]
  Day 8 (N=15, 16) | -3.11 (5.77) [-6.90 to -1.01] | -9.75 (9.88) [-12.18 to 1.06]
  Day 11 (N=16, 16) | -5.10 (5.07) [-7.34 to -0.78] | -5.51 (6.78) [-12.92 to -1.73]
  Day 15 (N=16, 16) | -0.49 (5.19) [-5.91 to 1.08] | -6.36 (9.79) [-15.92 to -0.21]
  Day 22 (N=14, 15) | -3.74 (7.28) [-8.25 to 0.00] | -4.26 (8.57) [-13.13 to 2.30]
  Day 29 (N=15, 16) | -1.17 (3.77) [-4.12 to 1.14] | -5.87 (12.34) [-9.62 to 3.00]
  Day 30 (N=15, 16) | -1.08 (3.64) [-2.08 to 1.01] | -2.17 (9.73) [-4.61 to 1.98]
  Day 31 (N=15, 16) | -1.03 (4.76) [-6.45 to 2.08] | -2.29 (10.16) [-6.17 to 3.71]
  Day 34 (N=15, 16) | 0.00 (6.07) [-3.92 to 2.94] | -2.85 (13.42) [-8.48 to 3.57]
  Day 36 (N=14, 16) | -1.08 (6.94) [-3.92 to 3.11] | -1.11 (7.39) [-6.55 to 2.18]
  Day 39 (N=16, 15) | -0.60 (5.15) [-4.60 to 2.66] | -1.93 (7.79) [-10.11 to 3.19]
  Day 43 (N=15, 15) | -1.04 (7.91) [-4.12 to 2.15] | -0.82 (6.78) [-9.27 to 2.96]
  Day 57 (N=15, 16) | -2.08 (5.52) [-6.86 to 2.27] | -1.64 (11.11) [-9.92 to 2.59]
  Day 71 (N=15, 16) | 2.06 (5.56) [-3.41 to 5.21] | -4.98 (9.38) [-15.07 to 1.88]
  Day 85 (N=14, 15) | 1.06 (6.37) [-6.86 to 4.55] | -6.87 (10.81) [-15.06 to 4.49]
  Day 113 (N=15, 16) | 0.00 (9.48) [-4.12 to 4.67] | -4.88 (7.94) [-8.71 to 1.12]

6. Secondary Outcome: Percent Change From Baseline in Serum Phosphorus Over Time
Time Frame: Baseline and Days 2, 3, 6, 8, 11, 15, 22, 29, 30, 31, 34, 36, 39, 43, 57, 71, 85, and 113
Population: Safety analysis set with available data at each time point
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Severe CKD | ESRD
Number analyzed (Participants) | 16 | 16
percent change
  Day 2 (N=16, 15) | -5.97 (10.42) [-12.14 to -2.41] | -20.00 (15.51) [-28.07 to -15.63]
  Day 3 (N=16, 15) | -10.37 (15.25) [-14.72 to -1.72] | -25.93 (24.26) [-35.71 to 2.27]
  Day 6 (N=16, 15) | -19.09 (15.81) [-25.47 to -8.22] | -24.56 (26.43) [-42.50 to -3.13]
  Day 8 (N=15, 16) | -13.46 (14.96) [-22.50 to -5.13] | -31.16 (35.81) [-40.92 to -7.81]
  Day 11 (N=16, 14) | -19.38 (10.93) [-26.14 to -12.86] | -33.29 (29.13) [-40.48 to -15.63]
  Day 15 (N=16, 16) | -10.00 (9.15) [-14.39 to -4.11] | -27.64 (26.62) [-40.00 to -16.75]
  Day 22 (N=15, 16) | -15.38 (17.27) [-28.21 to -3.57] | -25.89 (34.20) [-44.35 to -2.98]
  Day 29 (N=15, 16) | -5.13 (13.22) [-21.21 to 3.13] | -21.64 (22.06) [-27.50 to -10.00]
  Day 30 (N=15, 15) | -5.71 (13.63) [-20.51 to 3.45] | -31.25 (20.94) [-35.56 to -17.54]
  Day 31 (N=15, 15) | -7.14 (13.20) [-17.31 to 2.22] | -19.30 (20.69) [-22.50 to -9.38]
  Day 34 (N=15, 15) | -5.41 (14.23) [-15.38 to 3.57] | -15.00 (28.53) [-30.00 to 2.27]
  Day 36 (N=14, 16) | -4.84 (13.80) [-12.50 to 6.25] | -19.38 (18.77) [-36.61 to -11.00]
  Day 39 (N=16, 14) | -8.30 (11.72) [-14.45 to 0.94] | -18.89 (21.00) [-33.33 to 0.00]
  Day 43 (N=15, 15) | -6.82 (16.53) [-10.26 to 9.38] | -6.25 (30.76) [-40.48 to 7.50]
  Day 57 (N=15, 16) | -11.43 (11.65) [-21.15 to -3.45] | -7.18 (30.00) [-41.01 to 8.94]
  Day 71 (N=15, 16) | -3.45 (16.32) [-18.18 to 2.27] | -0.05 (45.15) [-30.95 to 32.50]
  Day 85 (N=15, 16) | -7.69 (14.51) [-25.64 to 3.13] | -6.04 (30.74) [-23.15 to 7.81]
  Day 113 (N=15, 16) | -7.14 (10.07) [-18.18 to 0.00] | -8.99 (33.92) [-19.87 to 25.00]

7. Secondary Outcome: Percent Change From Baseline in Serum Magnesium Over Time
Time Frame: Baseline and Days 2, 3, 6, 8, 11, 15, 22, 29, 30, 31, 34, 36, 39, 43, 57, 71, 85, and 113
Population: Safety analysis set with available data at each time point
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Severe CKD | ESRD
Number analyzed (Participants) | 16 | 16
percent change
  Day 2 (N=16, 15) | 0.00 (7.54) [-4.76 to 5.01] | -3.85 (7.47) [-7.41 to 4.55]
  Day 3 (N=16, 15) | 0.00 (10.94) [-5.26 to 8.20] | 0.00 (6.65) [-4.55 to 0.00]
  Day 6 (N=16, 15) | 2.50 (8.58) [-4.65 to 9.52] | 4.00 (14.39) [0.00 to 9.09]
  Day 8 (N=15, 16) | 4.76 (7.47) [-4.55 to 9.52] | 0.00 (10.46) [-8.15 to 4.55]
  Day 11 (N=16, 14) | 2.38 (10.29) [-4.77 to 10.53] | 0.00 (6.12) [-4.35 to 3.45]
  Day 15 (N=16, 16) | 0.00 (10.78) [-4.65 to 10.03] | 0.00 (7.88) [-4.76 to 2.27]
  Day 22 (N=15, 16) | 10.53 (9.14) [0.00 to 11.76] | 0.00 (9.24) [-2.00 to 4.45]
  Day 29 (N=15, 16) | 0.00 (9.87) [-4.76 to 4.76] | 2.27 (12.57) [-8.47 to 11.03]
  Day 30 (N=15, 15) | 0.00 (16.15) [-5.26 to 10.00] | -4.55 (8.87) [-13.64 to 0.00]
  Day 31 (N=15, 15) | 0.00 (12.46) [-5.26 to 5.88] | 0.00 (7.94) [-9.09 to 0.00]
  Day 34 (N=15, 15) | 0.00 (7.79) [-5.26 to 4.76] | 0.00 (7.85) [-6.90 to 5.26]
  Day 36 (N=14, 16) | 0.00 (9.79) [-5.88 to 4.76] | -4.45 (7.47) [-9.90 to 0.00]
  Day 39 (N=16, 14) | 0.00 (12.06) [-4.55 to 4.88] | -4.35 (8.68) [-13.64 to 0.00]
  Day 43 (N=15, 15) | 0.00 (8.31) [-4.76 to 5.88] | 3.45 (9.00) [-8.70 to 4.76]
  Day 57 (N=15, 16) | 5.00 (15.87) [0.00 to 9.52] | 0.00 (8.50) [-6.02 to 7.99]
  Day 71 (N=15, 16) | 0.00 (9.15) [-5.00 to 5.88] | 0.00 (11.74) [-8.19 to 9.52]
  Day 85 (N=15, 16) | 0.00 (9.21) [-9.09 to 5.88] | 4.12 (12.40) [-8.39 to 9.31]
  Day 113 (N=15, 16) | 0.00 (11.87) [-9.09 to 15.00] | 1.92 (9.46) [-4.45 to 8.55]

8. Secondary Outcome: Number of Participants With Adverse Events
Description: The severity of each adverse event (AE) was graded using the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0. The investigator assessed whether AEs were possibly related to study drug by answering the question: "Is there a reasonable possibility that the event may have been caused by the investigational product?" Abnormal laboratory findings without clinical significance (based on the investigator's judgment) were not recorded as AEs, however, laboratory value changes that required treatment or adjustment in current therapy were considered AEs. A serious adverse event is defined as an adverse event that meets at least 1 of the following serious criteria: • fatal, • life-threatening (places the participant at immediate risk of death), • requires in-patient hospitalization or prolongation of existing hospitalization, • results in persistent or significant disability/incapacity, • congenital anomaly/birth defect, and/or • other medically important serious event.
Time Frame: 113 days
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | Severe CKD | ESRD
Number analyzed (Participants) | 16 | 16
participants
  Any adverse event (AE) | 10 | 15
  Adverse events Grade >=3 | 3 | 7
  Serious adverse events | 1 | 2
  Leading to discontinuation of study drug | 0 | 0
  Leading to discontinuation from study | 0 | 0
  Fatal adverse events | 0 | 0
  Hypocalcemia adverse events | 3 | 10
  Hypomagnesemia adverse events | 0 | 0
  Hypophosphatemia adverse events | 0 | 1
  Treatment-related adverse events (TRAE) | 2 | 10
  Treatment-related adverse events Grade >=3 | 0 | 2
  Treatment-related serious adverse events | 0 | 0
  TRAE leading to discontinuation of study drug | 0 | 0
  TRAE leading to study discontinuation | 0 | 0

9. Secondary Outcome: Maximum Observed Serum Denosumab Concentration (Cmax)
Description: Serum concentrations of denosumab were measured by an enzyme-linked immunosorbent assay (ELISA). The lower limit of quantification (LLOQ) was 20 ng/mL.
Time Frame: Days 1 and 29 (predose), and on Days 8, 15, 36, 43, 57, 71, 85, and 113
Population: Pharmacokinetic (PK) Parameter Analysis Set (all participants who received at least 1 dose of denosumab and for whom PK parameter estimates could be derived)
Measure: Mean (Standard Deviation); unit: μg/mL
Groups:
- Severe CKD - Dose 1: Participants with severe CKD received 120 mg denosumab administered subcutaneously on Day 1.
- ESRD - Dose 1: Participants with ESRD requiring dialysis received 120 mg denosumab administered subcutaneously on Day 1.
- Severe CKD - Dose 2: Participants with severe CKD received 120 mg denosumab administered subcutaneously on Day 29.
- ESRD - Dose 2: Participants with ESRD requiring dialysis received 120 mg denosumab administered subcutaneously on Day 29.
Arm/Group | Severe CKD - Dose 1 | ESRD - Dose 1 | Severe CKD - Dose 2 | ESRD - Dose 2
Number analyzed (Participants) | 14 | 16 | 15 | 16
μg/mL | 10.5 (3.6) | 8.17 (4.22) | 16.1 (5.2) | 14.5 (7.4)

10. Secondary Outcome: Time to Maximum Observed Serum Denosumab Concentration (Tmax)
Description: as for outcome 9
Time Frame: Days 1 and 29 (predose), and on Days 8, 15, 36, 43, 57, 71, 85, and 113
Population: PK Parameter Analysis Set
Measure: Median (Full Range); unit: days
Arm/Group | Severe CKD - Dose 1 | ESRD - Dose 1 | Severe CKD - Dose 2 | ESRD - Dose 2
Number analyzed (Participants) | 14 | 16 | 15 | 16
days | 14 (3.6) [7.0 to 28] | 14 (4.22) [7.0 to 28] | 14 (5.2) [7.0 to 14] | 7.0 (7.4) [7.0 to 28]

11. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time 0 to 4 Weeks (AUC0-4wks) After Dose 1
Description: Estimated using the linear trapezoidal method.
Time Frame: Days 1, 8, 15, and 29 (predose)
Population: PK Parameter Analysis Set
Measure: Mean (Standard Deviation); unit: μg*day/mL
Arm/Group | Severe CKD - Dose 1 | ESRD - Dose 1
Number analyzed (Participants) | 14 | 16
μg*day/mL | 233 (75) | 177 (91)

12. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time 0 to 12 Weeks (AUC0-12wks) After Dose 2
Description: Estimated using the linear trapezoidal method.
Time Frame: Days 29 (predose), 36, 43, 57, 71, and 85
Population: PK Parameter Analysis Set
Measure: Mean (Standard Deviation); unit: μg*day/mL
Arm/Group | Severe CKD - Dose 2 | ESRD - Dose 2
Number analyzed (Participants) | 15 | 16
μg*day/mL | 853 (260) | 607 (262)

13. Secondary Outcome: Percent Change From Baseline in Serum C-Telopeptide Over Time
Time Frame: Baseline and Days 1 and 29 (predose), and on Days 8, 15, 36, 43, 57, 71, 85, and 113
Population: Pharmacodynamic Analysis Set (all participants who received at least 1 dose of denosumab and from whom baseline and at least 1 postbaseline value was collected)
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Severe CKD | ESRD
Number analyzed (Participants) | 16 | 16
percent change
  Day 8 (N=15, 16) | -63.0 (24.3) [-75.0 to -39.4] | -79.1 (13.6) [-87.8 to -68.8]
  Day 15 (N=16, 16) | -60.7 (23.6) [-73.0 to -38.3] | -79.3 (11.9) [-87.1 to -69.8]
  Day 29 (N=15, 16) | -58.4 (24.7) [-74.7 to -39.4] | -81.5 (12.3) [-87.0 to -67.8]
  Day 36 (N=15, 16) | -63.0 (24.2) [-75.0 to -39.4] | -79.4 (13.1) [-88.2 to -69.9]
  Day 43 (N=15, 15) | -58.4 (24.5) [-75.0 to -39.4] | -77.7 (13.4) [-87.0 to -69.3]
  Day 57 (N=15, 16) | -58.4 (24.0) [-75.0 to -39.4] | -81.7 (11.7) [-87.2 to -68.0]
  Day 71 (N=15, 16) | -58.4 (24.0) [-75.0 to -39.4] | -76.4 (13.8) [-87.9 to -68.2]
  Day 85 (N=15, 16) | -57.4 (24.0) [-75.0 to -39.4] | -75.9 (12.0) [-85.9 to -68.1]
  Day 113 (N=15, 16) | -50.2 [-75.0 to -39.4] | -75.6 [-88.5 to -63.3]

14. Secondary Outcome: Number of Participants Who Developed Anti-denosumab Antibodies
Time Frame: From Day 1 (predose) to Day 113
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | Severe CKD | ESRD
Number analyzed (Participants) | 16 | 16
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 113 days
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
  Summary of Adverse Events includes only those subjects who received at least one dose of investigational product.
  ESRD = End stage renal disease requiring dialysis.
Groups:
- Denosumab 120 mg - Severe: Participants with severe chronic kidney disease (CKD; defined as creatinine clearance < 30 mL/min) received two 120 mg doses of denosumab administered subcutaneously on Day 1 and Day 29.
- Denosumab 120 mg - ESRD: Participants with end-stage renal disease (ESRD) requiring dialysis received two 120 mg doses of denosumab administered subcutaneously on Day 1 and Day 29.
- Denosumab 120 mg - All Subjects: Participants received two 120 mg doses of denosumab administered subcutaneously on Day 1 and Day 29.
Arm/Group | Denosumab 120 mg - Severe | Denosumab 120 mg - ESRD | Denosumab 120 mg - All Subjects
Serious Adverse Events (participants affected / at risk) | 1/16 | 2/16 | 3/32
Other Adverse Events (participants affected / at risk) | 10/16 | 15/16 | 25/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Denosumab 120 mg - Severe (N=16) | Denosumab 120 mg - ESRD (N=16) | Denosumab 120 mg - All Subjects (N=32)
Ileitis (Gastrointestinal disorders) | 0 | 1 | 1
Asthenia (General disorders) | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Denosumab 120 mg - Severe (N=16) | Denosumab 120 mg - ESRD (N=16) | Denosumab 120 mg - All Subjects (N=32)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 1
Pericarditis (Cardiac disorders) | 0 | 1 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 1
Hearing impaired (Ear and labyrinth disorders) | 0 | 1 | 1
Hyperparathyroidism (Endocrine disorders) | 0 | 1 | 1
Hyperparathyroidism secondary (Endocrine disorders) | 1 | 1 | 2
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 3
Sensitivity of teeth (Gastrointestinal disorders) | 1 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 1
Sarcoidosis (Immune system disorders) | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1
Otitis media (Infections and infestations) | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 2
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 1 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 1
Vascular graft complication (Injury, poisoning and procedural complications) | 0 | 1 | 1
Blood calcium decreased (Investigations) | 1 | 0 | 1
Blood parathyroid hormone decreased (Investigations) | 1 | 0 | 1
Electrocardiogram PR shortened (Investigations) | 0 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 3 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 10 | 12
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Arterial stenosis (Vascular disorders) | 0 | 1 | 1
Hypertension (Vascular disorders) | 1 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.